CLINICAL TRIAL: NCT05314270
Title: Evaluation of Non-B Non-C Liver Cirrhosis in A EL-Rajhi Assuit University Hospital: A Retrospective-Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman mohammed abdelrahman morsi, Doctor, Assiut University
Other Study IDs: Non-B Non-C Liver cirrhosis
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Non-B Non-C Liver Cirrhosis
MeSH Terms: interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic tests — Diaagnostic tests for all pt diagnosed as Non-B Non-C Liver Cirrhosis
  Other Names: 24h copper in urine.. Iron profile.. Liver biopsy

SUMMARY:
To study the etiologies of patients diagnosed as non-B, non-C liver cirrhosis (NBNC-LC).

To describe the different patient's outcomes.

DETAILED DESCRIPTION:
Liver cirrhosis is the ultimate fate of many hepatic insults that may be viral, immunologic, and metabolic or even cryptogenic. (Tsochatzis EA et al., 2014)

Recently, Non-Alcoholic Fatty Liver Disease (NAFLD) present a serious health burden worldwide that affects around 25% of the global adult population with a prevalence of around 31.8% in the Middle East. (Younossi ZM, et al., 2019)

Most of Egyptian patients presented with end-stage liver disease are secondary to post-hepatitic cirrhosis is estimated to be more than 80% of cases. (Guerra J et al., 2012)

The real profile of non-B, non-C etiologies of liver cirrhosis, in Egyptian patients, is still not fully evaluated.

ELIGIBILITY:
Inclusion Criteria:

* All pateints diagnosed as Non-B Non-C Liver Cirrhosis in the period from 2017_2023

Exclusion Criteria:

* We will exclude the pateints that will be diagnosed as HBV-HCV induced Liver Cirrosis

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All pateints diagnosed as Non-B Non-C Liver Cirrhosis in the period from 2017_2023
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Detection of different etiologies of liver cirrhosis that not related to HBV or HCV in our community | Base line

SECONDARY OUTCOMES:
Detection of the most common etiologies of Non B Non C liver cirrhosis in our community | Baseline